CLINICAL TRIAL: NCT05444530
Title: A Phase 1 Study of VAC85135, a Neoantigen Vaccine Regimen, Concurrently Administered With Ipilimumab for the Treatment of Myeloproliferative Neoplasms
Brief Title: A Study of VAC85135, a Neoantigen Vaccine Regimen, Concurrently Administered With Ipilimumab for the Treatment of Myeloproliferative Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109149; VAC85135MPN1001 (Other: Janssen Research & Development, LLC); 2021-006033-20 (EudraCT Number); 2022-501913-30-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Myeloproliferative Neoplasms
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Participants with essential thrombocythemia (ET) and myelofibrosis (MF) will receive VAC85135 target dose intramuscular (IM) injection in the safety lead-in cohort (Cohort 0). Participants in subsequent cohorts will receive VAC85135 target dose IM injection along with ipilimumab intravenous (IV) infusion. Ipilimumab dose may be escalated based on dose limiting toxicity (DLT) observations.
  Interventions: Biological: VAC85135; Drug: Ipilimumab
- Dose Expansion (Experimental): Participants with polycythemia vera (PV) or post-polycythemia vera myelofibrosis, ET and MF will receive VAC85135 target dose IM injection with ipilimumab IV infusion at the dose(s) determined by study evaluation team (SET).
  Interventions: Biological: VAC85135; Drug: Ipilimumab

INTERVENTIONS:
Biological: VAC85135 — Participants will receive VAC85135 as IM injection.
Drug: Ipilimumab — Participants will receive Ipilimumab as IV infusion.

SUMMARY:
The purpose of this study is to evaluate the safety of VAC85135 administered with ipilimumab for the treatment of myeloproliferative neoplasms (MPNs).

ELIGIBILITY:
Inclusion Criteria:

* Be positive for a CALR (calreticulin) mutation: Type 1 or Type 2; Type 1-like, or Type 2-like may be considered with Sponsor approval; or positive for the JAK2V617F (Janus kinase 2 with valine 617 to phenylalanine mutation) mutation with HLA-A02:01 (human leukocyte antigens) per medical history or local testing
* Have an Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1 or 2
* Have the following hematologic laboratory values: Leukocytes greater than or equal to (>=) 1.5*10^9 per liter, Neutrophils >=1.0*10^9 per liter, Platelets >=20*10^9 per liter, Hemoglobin greater than (>) 7 gram per deciliter (g/dL)
* Have the following chemistry laboratory values: Alanine aminotransferase (ALT): less than or equal to (<=) 3*upper limit of normal (ULN), Aspartate aminotransferase (AST): <=3*ULN, Total bilirubin: <=1.5*ULN, and glomerular filtration rate >=40 milliliter per minute (mL/min)
* A female participant of childbearing potential must agree to all the following during the study and for 6 months after the last dose of study treatment: use a barrier method of contraception, use a highly effective preferably user-independent method of contraception, not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction, not plan to become pregnant, not to breast-feed
* A male participant must agree to all the following during the study and for 90 days after the last dose of study treatment: wear a condom when engaging in any activity that allows for passage of ejaculate to another person, not to father a child, not to donate sperm or freeze for future use for the purpose of reproduction

Exclusion Criteria:

* History of any significant medical condition per investigators judgment (example: severe asthma/chronic obstructive pulmonary disease (COPD), poorly regulated heart condition, insulin dependent diabetes mellitus)
* Serious known clinically relevant allergies or earlier anaphylactic reactions
* Currently pregnant or breastfeeding
* Prior treatment with any Janus kinase 1/2 (JAK1/2) inhibitor
* Known sensitivity or contraindications to the use of Ipilimumab per local prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicity (DLT) | Baseline (Day 1) up to Day 78
  Number of participants with a DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity. Toxicities will be graded for severity according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 79 weeks
  Number of participants with AEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical product. AEs will be graded as Grade 1: Mild- asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate- minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL); Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4- Life-threatening consequences- urgent intervention indicated; Grade 5: Death related to AE.

SECONDARY OUTCOMES:
Number of Participants With Antigen-specific T-cell response | Up to end of treatment (EOT) (Up to 64 weeks)
  Number of participants with antigen-specific T-cell response will be reported.
Number of Participants With Overall Response per Revised Response Criteria by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) Consensus Report | Up to 79 weeks
  Overall response will be measured by complete remission, partial remission, clinical improvement, anemia response, spleen response, symptoms response, progressive disease, stable disease and relapse as per the revised IWG-MRT and ELN response criteria for myelofibrosis (MF).
Number of Participants Disease Response at Weeks 24, 48 and End of Treatment (EOT) per Modified IWG-MRT Criteria | Weeks 24, 48 and EOT (64 weeks)
  Number of participants with disease response as per the modified IWG-MRT criteria will be reported.
Number of Participants With Peripheral Blood Mutant Calreticulin (mutCALR) and Janus Kinase 2 With V617F Mutation (JAK2V617F) Allele Burden | Up to end of treatment (EOT) (Up to 64 weeks)
  Number of participants with peripheral blood mutCALR and JAK2V617F allele burden will be reported.
Number of Participants With Transfusion Burden | Up to end of treatment (EOT) (Up to 64 weeks)
  Number of participants with transfusion burden will be reported.
Number of Participants With Patient-reported Symptoms on Therapy | Up to end of treatment (EOT) (Up to 64 weeks)
  Number of participants with patient-reported symptoms on therapy will be reported.
Time to Progression of Myeloproliferative Neoplasms (MPNs) | Up to end of treatment (EOT) (Up to 64 weeks)
  Time to progression of MPNs (polycythemiavera [PV], essential thrombocythemia [ET], and primary myelofibrosis [PMF]) will be reported.
Time to Initiation of Next Therapy | Up to 79 weeks
  Time to initiation of next therapy for myeloproliferative neoplasms (MPNs) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- United States (4):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- United Kingdom (3):
  - Guy's and St Thomas' Hospital, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency